CLINICAL TRIAL: NCT04420676
Title: Synbiotic Therapy of Gastrointestinal Symptoms During Covid-19 Infection: A Randomized, Double-blind, Placebo Controlled, Telemedicine Study (SynCov Study)
Brief Title: Synbiotic Therapy of Gastrointestinal Symptoms During Covid-19 Infection
Acronym: SynCov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SynCov
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: COVID

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Group 1: receiving a probiotic mixture (Omni-Biotic® 10 AAD) twice a day
  Interventions: Dietary Supplement: Omnibiotic AAD
- Placebo (Placebo Comparator): Group 2: receiving a similar looking and tasting placebo without bacteria twice a day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omnibiotic AAD — Bacterial strains in Omni-Biotic® 10 AAD are Bifidobacterium bifidum W23, Bifidobacterium lactis W51, Enterococcus faecium W54, Lactobacillus acidophilus W37, Lactobacillus acidophilus W55, Lactobacillus paracasei W20, Lactobacillus plantarum W1, Lactobacillus plantarum W62, Lactobacillus rhamnosus W71 and Lactobacillus salivarius W24 which are embedded in a matrix containing maize starch, maltodextrin, inulin, potassium chloride, hydrolysed rice protein, magnesium sulphate, fructooligosaccharide (FOS), enzymes (amylases), vanilla flavour and manganese sulphate
  Other Names: Ecologic AAD
  Arms: Probiotic
Dietary Supplement: Placebo — matrix containing maize starch, maltodextrin, inulin, potassium chloride, hydrolysed rice protein, magnesium sulphate, fructooligosaccharide (FOS), enzymes (amylases), vanilla flavour and manganese sulphate.
  Arms: Placebo

SUMMARY:
We hypothesize that the intake of Omni-Biotic® 10 AAD can reduce intestinal inflammation and improves dysbiosis in Covid-19 disease. We further hypothesize that Omni-Biotic® 10 AAD can reduce the duration of diarrhea, stool frequency, improve stool consistency, improve other gastrointestinal symptoms of Covid-19, reduce disease duration and severity.

The investigators aim to perform a randomized, double blind, placebo-controlled study using telemedicine in patients with Covid-19 disease.

DETAILED DESCRIPTION:
The outbreak of the novel coronavirus (SARS-CoV-2)-infected disease (COVID-19) began in Wuhan, Hubei province in December 2019, spread throughout China in early 2020 and developed as a pandemic thereafter. Although the virus mainly causes respiratory symptoms, GI (gastrointestinal) presentations have been reported in and outside of China. Patients may present with anorexia, nausea, vomiting, diarrhea and abdominal discomfort. Also, faecal-oral transmission of the virus is currently discussed. Preliminary, unpublished data from China suggest that patients with GI symptoms may suffer more frequently from severe courses of the disease. Clinical studies show an incidence rate of diarrhea ranging from 2% to 50% of cases. It may precede or trail respiratory symptoms. A pooled analysis revealed an overall percentage of diarrhea onset of 10.4%. SARS-CoV-2 uses the angiotensin-converting enzyme 2 (ACE2) for cellular entry. ACE2 is expressed in the small intestinal epithelia as well as in the upper esophagus, liver, and colon. SARS-CoV-2 binding affinity to ACE2 is significantly higher (10-20 times) compared with SARS-CoV. Diarrhea is associated with prolonged symptoms and viral carriage.

Clinical information on the characteristics of Covid-19 diarrhea is scarce. The duration of diarrhea is around 4 days with 3-4 loose stools per day. Faecal calprotectin is elevated in stool of patients with Covid-19 diarrhea, indicating a relation between gastrointestinal symptoms and this well-established inflammation biomarker.

So far, no therapy is available for Covid-19 infection in general or for Covid-19 induced diarrhea. Rehydration and potassium monitoring should be performed as in all patients with diarrhea. It is important to underline that antivirals and antibiotics are often used for COVID-19 treatment or treatment of bacterial superinfections, involving a likely alteration of the gut microbiota and causing diarrhea. It is therefore plausible that the gut microbiota could be a new therapeutic target and that probiotics or synbiotics (combination of probiotics with prebiotics) could have a role in the management of these patients. The China's National Health Commission recommended the use of probiotics for the treatment of patients with severe COVID-19 in order to preserve intestinal balance and to prevent secondary bacterial infections without any available clinical studies to support this and probiotics apparently were used in Zhejiang during the Covid-19 pandemic. Although there is no specific data on the effects of probiotics on SARS-CoV2 infections, meta-analyses show that probiotics are effective in the treatment of upper respiratory tract infections and viral gastroenteritis of other origins. Furthermore, Enterococcus faecium has been shown to have antiviral effects in enteropathogenic coronavirus transmissible gastroenteritis virus infections in piglets. We therefore aim to assess the role of synbiotics in the therapy of Covid-19 infection with gastrointestinal symptoms.

ELIGIBILITY:
Inclusion criteria

* 18 years or older
* Covid-19 infection diagnosed by a positive SARS-Cov-2 PCR (Polymerase chain reaction) result from a nasopharyngeal swab
* Informed (tele)consent Exclusion criteria
* Pre-existing diarrhoea (including but not restricted to chronic inflammatory bowel disease, chronic diarrhea of other causes, acute diarrheal illness -4 to -1 week before inclusion)
* Antibiotic therapy -4 to -1 week before inclusion
* Probiotic treatment -4 to -1 week before inclusion
* Technical difficulties to perform telemedicine study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stool calprotectin | 30 days
  measured by ELISA

SECONDARY OUTCOMES:
Stool frequency | 30 days
  stool evacuations per days
Stool consistency | 30 days
  Stool consistency according to Bristol stool scale for each evacuation, score 1-7, a higher score means a lower stool consistancy
Gastrointestinal symptoms | 30 days
  presence of anorexia, nausea, vomiting, abdominal pain, bloating (yes/no)
Duration of Covid-19 disease | 30 days
  days patients feel sick, are not able to work or are on sick leave
Severity of Covid-19 disease | 30 days
  mild/moderate/severe
Diarrhea | 30 days
  3 or more stool evacuations, consistency Bristol stool scale 5-7
Stool Zonulin | 30 days
  measured by ELISA
Microbiome composition | 30 days
  16S RNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
Upload of microbiome sequences and metadata to a repository
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after completion
Access Criteria: free